CLINICAL TRIAL: NCT00179309
Title: A Randomized Pilot Phase II Study of Docetaxel Alone or in Combination With PANVAC(Trademark)-V (Vaccinia) and PANVAC(Trademark)-F (Fowlpox) in Adults With Metastatic Breast Cancer
Brief Title: Docetaxel Alone or in Combination With Vaccine to Treat Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, James Gulley, M.D., Principal investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 050229; 05-C-0229; NCT00217750 (obsolete NCT alias)
Record Dates: First submitted 2005-09-15; First posted 2005-09-15 (Estimated); Results first posted 2013-06-27 (Estimated); Last update posted 2014-07-15 (Estimated); Status verified 2014-06

CONDITIONS: Breast Cancer
Keywords: CEA; MUC-1; Immunotherapy; GM-CSF; Vaccine; Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I - PANVAC + docetaxel (Experimental): Patients receive vaccinia-carcinoembryonic antigen (CEA)- mucin-1 (MUC-1)- triad of costimulatory molecules (TRICOM) vaccine subcutaneously (SC) once and sargramostim, or granulocyte macrophage colony stimulating factor (GM-CSF) SC once daily for 4 days in week -2. Patients also receive fowlpox-CEA-MUC-1-TRICOM vaccine SC once and GM-CSF SC once daily for 4 days in weeks 1, 5, and 9. Patients also receive docetaxel intravenous (IV) over 30 minutes once weekly in weeks 1-3, 5-7, and 9-11. After week 12, patients with no disease progression continue with docetaxel once weekly for 3 weeks followed by 1 week of rest and fowlpox-CEA-MUC-1-TRICOM vaccine plus GM-CSF every 4 weeks until disease progression.
  Interventions: Drug: Docetaxel; Biological: PANVAC-V; Biological: PANVAC-F; Biological: Sargramostim
- Arm II - Docetaxel alone (Experimental): Patients receive docetaxel as in arm I. After week 12, patients with disease progression discontinue docetaxel and receive vaccinia-carcinoembryonic antigen (CEA)- mucin 1(MUC-1)-triad of costimulatory molecules (TRICOM) vaccine, fowlpox-CEA-MUC-1-TRICOM vaccine, and sargramostim, or granulocyte macrophage colony stimulating factor (GM-CSF) as in arm I until further disease progression. Patients with no disease progression after week 12 continue with docetaxel as in arm I until disease progression.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — 35 mg/m^2 intravenous 30-60 minutes once a week for 3 consecutive weeks with 1 week off drug.
  Other Names: Taxotere
Biological: PANVAC-V — 2 x 10^8 PFU
  Arms: Arm I - PANVAC + docetaxel
Biological: PANVAC-F — 1 x 10^9 PFU
  Arms: Arm I - PANVAC + docetaxel
Biological: Sargramostim — Given subcutaneously under the skin, usually in the thigh on the day of vaccination and daily for the next 3 days.
  Other Names: GM-CSF
  Arms: Arm I - PANVAC + docetaxel

SUMMARY:
This study will test whether giving a combination of a vaccine together with docetaxel is more effective against breast cancer than docetaxel alone. The Food and Drug Administration has approved docetaxel to treat many cancers, including breast cancer. The vaccine consists of three parts: 1) a "priming vaccine" called PANVAC (PAN (all) VAC (vaccine)) trademark [TM]-V, which is made from vaccinia virus; 2) a "boosting vaccine" called PANVAC[TM]-F, made from fowlpox virus; and 3) sargramostim, or granulocyte macrophage colony stimulating factor (GM-CSF), a protein that may help boost the immune system. Human genes are inserted into the vaccinia and fowlpox viruses to cause production of carcinoembryonic antigen (CEA) and mucin 1 (MUC-1)-two proteins that are often produced by cancer cells and can be used as a target for the immune system to attack the cancer. Another type of deoxyribonucleic acid (DNA) is inserted to cause production of other proteins that enhance immune activity.

Patients 18 years of age or older with metastatic breast cancer (disease that has spread beyond the original site) and whose cancer produces CEA or mucin 1 (MUC-1) protein may be eligible for this study. Patients must have antigen type human leukocyte antigen A2 (HLA-A2). They may have received adjuvant docetaxel treatment at least 3 months before entering this study, prior hormonal therapy and up to three chemotherapy regimens. Candidates are screened with a medical history and physical examination, blood and urine tests, electrocardiogram, and computerized tomography (CT) or magnetic resonance imaging scans.

Participants are randomly assigned to one of two treatment groups - docetaxel alone or docetaxel plus vaccine - as follows:

Docetaxel Alone

All patients receive docetaxel. The drug is infused through a vein over 30 to 60 minutes once a week for 3 consecutive weeks with 1 week off drug. Patients also take dexamethasone 12 hours and 1 hour before and 12 hours after the docetaxel to help prevent fluid retention (edema) that docetaxel may cause.

Docetaxel Plus Vaccine

Participants receive the priming vaccination followed by monthly boosting vaccinations, along with the weekly docetaxel therapy. With every vaccination, patients also receive an injection of sargramostim to increase the number of immune cells at the vaccination site. Sargramostim injections are given the day of vaccination and daily for the next 3 days. All vaccine and sargramostim doses are given as injections under the skin, usually in the thigh. Patients are observed in the clinic for 1 hour after each injection.

Patients have blood tests every four weeks to monitor drug side effects and before every vaccination to check blood counts. A bone scan or CT scan (or both) is done every 2 to 3 months to check the response to treatment.

Patients may continue receiving treatment as long as their disease does not worsen and they can tolerate the treatment without significant side effects. Patients assigned to receive docetaxel alone whose disease progresses after 3 months on the drug may choose to receive the vaccine or come off the study to receive other treatment options. Patients are monitored with yearly telephone calls for up to 15 years.

DETAILED DESCRIPTION:
Background:

Weekly docetaxel therapy is currently used as a standard treatment for patients with metastatic breast cancer.

Although many patients initially respond to this form of therapy, the majority will eventually develop disease progression and die from their disease.

We have explored the use of combining pox vector vaccines with docetaxel. In a recent clinical trial, men with prostate cancer were given both the vaccine and docetaxel without any significant toxicity and the docetaxel did not diminish immune responses to the vaccine.

Objectives:

To evaluate progression free survival comparing PANVAC + docetaxel vs. docetaxel alone in patients with metastatic breast cancer.

To evaluate overall survival comparing PANVAC + docetaxel vs. docetaxel alone in patients with metastatic breast cancer.

To evaluate in both arms cluster of differentiation 8 (CD8+) T cell responses directed against carcinoembryonic antigen (CEA) and mucin (MUC-1) in human leukocyte antigen 2 (HLA-A2), A3, and A24 positive patients by interferon-gamma enzyme linked immunosorbent spot (ELISPOT) assay.

Eligibility:

Metastatic breast cancer (either male or female) with evidence of metastatic disease (must have radiographic evidence of disease) and life expectancy of at least 4 months.

Patients may have received unlimited prior hormonal therapy or chemotherapy, but no prior docetaxel for metastatic disease.

Hematological eligibility parameters within 16 days of starting therapy:

Granulocyte count greater than or equal to 1,500/mm^3, Platelet count greater than or equal to 100,000/mm^3, hemoglobin (Hgb) greater than or equal to 8 Gm/dL.

Design:

A randomized Phase II study evaluating the role of combining docetaxel with PANVAC[TM]-V (recombinant vaccinia containing the genes encoding for CEA, MUC-1, lymphocyte function-associated antigen 3 (LFA-3), intercellular adhesion molecule 1 (ICAM-1) and B7.1) and PANVAC[TM]-F (recombinant fowlpox containing the genes encoding for CEA, MUC-1, LFA-3, ICAM-1 and B7.1) vs. docetaxel alone to determine if the addition of the vaccine can prolong the time to disease progression as well as overall survival in patients with metastatic breast cancer.

Patients randomized to docetaxel alone may receive sequential therapy with PANVAC[TM]-V and PANVAC[TM]-F at time of disease progression.

In patients randomized to the concurrent therapy, PANVAC[TM]-V will be administered to patients 3 weeks prior to the start of chemotherapy as the initial vaccine.

The immune responses to CEA and MUC-1 will then be boosted by administration of PANVAC[TM]-F.

Sargramostim or granulocyte macrophage colony stimulating factor (GM-CSF) will be administered with each vaccine inoculation for four consecutive days only for patients treated at the National cancer Institute (NCI).

ELIGIBILITY:
* INCLUSION CRITERIA:
* Metastatic Breast Cancer (either male or female) with evidence of metastatic disease (must have radiographic evidence of measurable disease) on computed tomography (CT) scan or X-ray, or evidence of evaluable disease on bone scan that is consistent with metastasis and a life expectancy of at least 4 months. Patients may have received unlimited prior hormonal therapy and chemotherapy.
* Histologically confirmed adenocarcinoma of the breast cancer confirmed in the Pathology Clinical Center at National Cancer Institute (NCI), (or National Naval Medical Center (NNMC)) or MD Anderson Pathology Department prior to starting this study. Note: However, if no pathologic specimen is available, patients may enroll with a clinical course consistent with breast cancer and a pathological documentation of the disease.
* 18 years of age or greater.
* May have received docetaxel in the adjuvant setting at least 12 months prior to study entry.
* Able to understand and give informed consent.
* Able to avoid close household contact (close household contacts are those who share housing or have close physical contact) for at least two weeks after recombinant vaccinia vaccination with persons with active or a history of eczema or other eczematoid skin disorders; those with other acute, chronic or exfoliative skin conditions (e.g., atopic dermatitis, burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds) until condition resolves; pregnant or nursing women; children 3 years of age and under; and immunodeficient or immunosuppressed persons (by disease or therapy), including human immunodeficiency virus (HIV) infection. We have vaccinated over 700 cancer patients and have reported no cases of either self inoculation or person to person transmission of the virus.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1.
* Serum creatinine less than 1.5 times upper limits of normal (ULN) OR creatinine clearance on a 24 hour urine collection of greater than or equal to 60 mL/min, standard liver function tests (LFT) limitations for patients receiving docetaxel therapy include bilirubin within ULN and serum glutamic oxaloacetic transaminase (SGOT)/serum glutamic pyruvic transaminase (SGPT) less than 1.5 times the ULN. If transaminases are greater than 1.5 times the ULN up to 2 times the ULN (as currently indicated), then alk phos should be less than 2.5 times the ULN. (Patients with renal abnormalities should be evaluated for creatinine clearance (CrCl) and interstitial abnormalities. A Cr Cl of greater than or equal to 60ml/min measured or calculated and proteinuria less than 1000mg per 24 hours are eligible unless explained by non-renal causes.)
* Recovered completely from any grade 3 or 4 reversible hematologic and non hematologic toxicity associated with recent therapy. Typically this is 3-4 weeks for patients who most recently received cytotoxic therapy. Patients previously treated with mitomycin c or carboplatin will require a minimum of 6 weeks.
* Hematological eligibility parameters (within 16 days of starting therapy):

  1. Granulocyte count greater than or equal to1,500/mm^3
  2. Platelet count greater than or equal to 100,000/mm^3
  3. Hemoglobin (Hgb) greater than or equal to 8 Gm/dL
* Must agree to use effective birth control or abstinence during and for a period of 4 months after the last vaccination therapy.
* Patients whose tumors are estrogen receptor (ER) positive should have failed primary hormone therapy unless clinically indicated, i.e. in patients with visceral disease or symptomatic bone disease where up front chemotherapy is warranted. Patients who progressed or recurred following Trastuzumab (Herceptin) therapy if a patient is fluorescence in situ hybridization (FISH) positive or immunohistochemistry (IHC) 3+ positive for human epidermal growth factor receptor 2 (Her-2 neu). Those patients who have progressed on trastuzumab may continue to receive the drug by their referring physician. However, if trastuzumab has been discontinued at the time of enrolling on study, it cannot be resumed while a patient remains on study.
* Patients randomized to docetaxel alone (arm B) may at time of progression go on to receive vaccine alone if their ECOG performance status remains 0-1, and they do not have any uncontrolled pain or organ dysfunction that would require another intervention such as radiation or chemotherapy.

Furthermore, patients initially randomized to arm B that would like to cross over and continue vaccine therapy must meet on-study eligibility and exclusion criteria with the exception of liver transaminase requirement. Patients with liver transaminase levels within Grade 1 by Common Terminology Criteria for Adverse Events (CTCAE) v4.0 (up to 3 x ULN) will be allowed to crossover to vaccine.

* Patients should appear clinically stable (in the opinion of the principle investigator) to complete the full 3 month course of vaccination with an anticipated survival of 6 months or longer.
* No other active malignancies within the past 12 months (with the exception of non-melanoma skin cancers or carcinoma in situ of the bladder) or life threatening illnesses.
* Patients with cardiovascular symptoms should be fully evaluated for signs and symptoms of cardiovascular disease and other standard evaluations including electrocardiogram (EKG), chest X-ray, cardiac enzymes, and echocardiogram as clinically indicated.

EXCLUSION CRITERIA:

* Patients should have no evidence of being immunocompromised as listed below.

  1. Human immunodeficiency virus positivity due to the potential for decreased tolerance and risk for severe side effects
  2. Active autoimmune diseases requiring treatment or a history of autoimmune disease that might be stimulated by vaccine treatment. This requirement is due to the potential risks of exacerbating autoimmunity Patients with endocrine disease that is controlled by replacement therapy including thyroid disease and adrenal disease and vitiligo may be enrolled
  3. Concurrent use of systemic steroids, except for local (topical, nasal, or inhaled) steroid use
* History of allergy or untoward reaction to prior vaccination with vaccinia virus.
* Pregnant or breast-feeding women
* Altered immune function, including immunodeficiency or history of immunodeficiency; eczema; history of eczema, or other eczematoid skin disorders; or those with acute, chronic or exfoliative skin conditions (e.g. atopic dermatitis, burns, impetigo, varicella zoster, severe acne, or other open rashes or wounds)
* Serious intercurrent medical illness which would interfere with the ability of the patient to carry out the treatment program, including, but not limited to, inflammatory bowel disease, Crohn's disease, ulcerative colitis, or active diverticulitis
* Clinically active brain metastasis, or a history of seizures that have been active within one year
* Medical conditions, which, in the opinion of the investigators would jeopardize the patient or the integrity of the data obtained
* Prior docetaxel chemotherapy for metastatic disease
* Serious hypersensitivity reaction to egg products
* Clinically significant cardiomyopathy requiring treatment
* Chronic hepatitis infection, including B and C, because of potential immune impairment
* Although topical steroids are allowed, steroid eye-drops are contraindicated
* Patients who have received prior PANVAC vaccine therapy
* Patients with a prior history of allergy to eggs or egg products should not receive the vaccine
* Patients with cardiac disease that have fatigue, palpitation, dyspnea or angina with ordinary physical activity (New York Heart Association class 2 or greater) are not eligible.
* Prior splenectomy.
* Cardiac complications, including recent myocardial infarction or cerebrovascular accident within one year, and/or unstable or uncontrolled angina.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-09; Primary Completion 2013-02 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James L Gulley, M.D., Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - U.T.M.D. Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Background] Garnett CT, Schlom J, Hodge JW. Combination of docetaxel and recombinant vaccine enhances T-cell responses and antitumor activity: effects of docetaxel on immune enhancement. Clin Cancer Res. 2008 Jun 1;14(11):3536-44. doi: 10.1158/1078-0432.CCR-07-4025. PMID 18519787
- [Background] Gulley JL, Madan RA, Arlen PM. Enhancing efficacy of therapeutic vaccinations by combination with other modalities. Vaccine. 2007 Sep 27;25 Suppl 2(Suppl 2):B89-96. doi: 10.1016/j.vaccine.2007.04.091. Epub 2007 Jun 4. PMID 17573164
- [Background] Arlen PM, Pazdur M, Skarupa L, Rauckhorst M, Gulley JL. A randomized phase II study of docetaxel alone or in combination with PANVAC-V (vaccinia) and PANVAC-F (fowlpox) in patients with metastatic breast cancer (NCI 05-C-0229). Clin Breast Cancer. 2006 Jun;7(2):176-9. doi: 10.3816/CBC.2006.n.032. No abstract available. PMID 16800982
- [Background] Huang J, Jochems C, Talaie T, Anderson A, Jales A, Tsang KY, Madan RA, Gulley JL, Schlom J. Elevated serum soluble CD40 ligand in cancer patients may play an immunosuppressive role. Blood. 2012 Oct 11;120(15):3030-8. doi: 10.1182/blood-2012-05-427799. Epub 2012 Aug 28. PMID 22932804
- [Derived] Gorodetska I, Samusieva A, Lahuta T, Ponomarova O, Socha O, Kozeretska I. Exploring New Frontiers: Alternative Breast Cancer Treatments Through Glycocalyx Research. Breast J. 2025 May 22;2025:9952727. doi: 10.1155/tbj/9952727. eCollection 2025. PMID 40443562
- [Derived] Heery CR, Ibrahim NK, Arlen PM, Mohebtash M, Murray JL, Koenig K, Madan RA, McMahon S, Marte JL, Steinberg SM, Donahue RN, Grenga I, Jochems C, Farsaci B, Folio LR, Schlom J, Gulley JL. Docetaxel Alone or in Combination With a Therapeutic Cancer Vaccine (PANVAC) in Patients With Metastatic Breast Cancer: A Randomized Clinical Trial. JAMA Oncol. 2015 Nov;1(8):1087-95. doi: 10.1001/jamaoncol.2015.2736. PMID 26291768
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2005-C-0229.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Crossover was allowed so that patients randomized to B could receive the vaccine upon progression.
Groups:
- Arm I - PANVAC + Docetaxel: Patients receive vaccinia-carcinoembryonic antigen (CEA)- mucin-1 (MUC-1)- triad of costimulatory molecules (TRICOM) vaccine subcutaneously (SC) once and sargramostim, or granulocyte macrophage colony stimulating factor (GM-CSF) SC once daily for 4 days in week -2. Patients also receive fowlpox-CEA-MUC-1-TRICOM vaccine SC once and GM-CSF SC once daily for 4 days in weeks 1, 5, and 9. Patients also receive docetaxel intravenous (IV) over 30 minutes once weekly in weeks 1-3, 5-7, and 9-11. After week 12, patients with no disease progression continue with docetaxel once weekly for 3 weeks followed by 1 week of rest and fowlpox-CEA-MUC-1-TRICOM vaccine plus GM-CSF every 4 weeks until disease progression.
  PANVAC-V: given subcutaneously
  Sargramostim : given subcutaneously (NCI subjects only)
  PANVAC-F : given subcutaneously
  Docetaxel : given IV
- Arm II - Docetaxel Alone: Patients receive docetaxel as in arm I. After week 12, patients with disease progression discontinue docetaxel and receive vaccinia-carcinoembryonic antigen (CEA)- mucin 1(MUC-1)-triad of costimulatory molecules (TRICOM) vaccine, fowlpox-CEA-MUC-1-TRICOM vaccine, and sargramostim, or granulocyte macrophage colony stimulating factor (GM-CSF) as in arm I until further disease progression. Patients with no disease progression after week 12 continue with docetaxel as in arm I until disease progression.
  Docetaxel : given intravenous (IV)
Period: Treatment
Arm/Group | Arm I - PANVAC + Docetaxel | Arm II - Docetaxel Alone
Started | 25 | 23
Completed | 21 | 18
Not Completed | 4 | 5
Not completed — Toxicity | 2 | 3
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Allergy | 1 | 0
Period: Crossover
Arm/Group | Arm I - PANVAC + Docetaxel | Arm II - Docetaxel Alone
Started | 0 | 3 (Crossover was allowed so that patients randomized to B could receive the vaccine upon progression.)
Completed | 0 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm I - PANVAC + Docetaxel: Patients receive vaccinia-carcinoembryonic antigen (CEA)- mucin-1 (MUC-1)- triad of costimulatory molecules (TRICOM) vaccine subcutaneously (SC) once and sargramostim, or granulocyte macrophage colony stimulating factor (GM-CSF) SC once daily for 4 days in week -2. Patients also receive fowlpox-CEA-MUC-1-TRICOM vaccine SC once and GM-CSF SC once daily for 4 days in weeks 1, 5, and 9. Patients also receive docetaxel intravenous (IV) over 30 minutes once weekly in weeks 1-3, 5-7, and 9-11. After week 12, patients with no disease progression continue with docetaxel once weekly for 3 weeks followed by 1 week of rest and fowlpox-CEA-MUC-1-TRICOM vaccine plus GM-CSF every 4 weeks until disease progression.
  PANVAC-V : given subcutaneously
  Sargramostim : given subcutaneously (NCI subjects only)
  PANVAC-F : given subcutaneously
  Docetaxel : given IV
- Arm II - Docetaxel Alone: Patients receive docetaxel as in arm I. After week 12, patients with disease progression discontinue docetaxel and receive vaccinia-carcinoembryonic antigen (CEA)- mucin (MUC-1)-triad of costimulatory molecules (TRICOM) vaccine, fowlpox-CEA-MUC-1-TRICOM vaccine, and sargramostim, or granulocyte macrophage colony stimulating factor(GM-CSF) as in arm I until further disease progression. Patients with no disease progression after week 12 continue with docetaxel as in arm I until disease progression.
  Docetaxel : given intravenous (IV)
- Total: Total of all reporting groups
Arm/Group | Arm I - PANVAC + Docetaxel | Arm II - Docetaxel Alone | Total
Number analyzed (Participants) | 25 | 23 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 18 | 38
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.52 (10.52) | 53.01 (12.22) | 54.31 (11.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 22 | 47
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 25 | 20 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 3 | 10
  White | 17 | 18 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 23 | 48

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: Time between the first day of treatment and disease progression. Progression is assessed by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria. Progressive disease is a minimum of 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum of the longest diameter recorded since the treatment started or the appearance of one or more new measurable lesions.
Time Frame: 19.7 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I - PANVAC + Docetaxel | Arm II - Docetaxel Alone
Number analyzed (Participants) | 25 | 23
Months | 6.6 [3.7 to 9.4] | 3.8 [2.6 to 8.4]
Statistical Analysis 1: Comparison: Arm I - PANVAC + Docetaxel; 48 evaluable pts will be randomized in a 1:1 ratio between two arms (24 evaluable pts per arm). Using standard formulae (e.g. nQuery Advisor v5), this number was selected to provide 80% power to detect a difference between 4.2 month median progression free survival (PFS) on the docetaxel alone arm and 8 month median PFS on the arm receiving PANVAC plus docetaxel, with a one-tailed alpha=0.10,assuming 36 months accrual and an additional 12 months of follow-up after the last pt has been enrolled; Test type: Superiority or Other; p = 0.12, Log Rank — Multiple comparisons were not done

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 80 months
Measure: Number; unit: Participants
Arm/Group | Arm I - PANVAC + Docetaxel | Arm II - Docetaxel Alone
Number analyzed (Participants) | 25 | 23
Participants | 23 | 23

ADVERSE EVENTS:
Arm/Group | Arm I - PANVAC + Docetaxel | Arm II - Docetaxel Alone
Serious Adverse Events (participants affected / at risk) | 3/25 | 2/23
Other Adverse Events (participants affected / at risk) | 23/25 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - PANVAC + Docetaxel (N=25) | Arm II - Docetaxel Alone (N=23)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify -stomatitis) (Gastrointestinal disorders) | 0 (0) | 1 (2)
Nervous system disorders - Other, specify -neuropathy, hands and feet (Nervous system disorders) | 0 (0) | 1 (1)
Vascular access complication (Vascular disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I - PANVAC + Docetaxel (N=25) | Arm II - Docetaxel Alone (N=23)
Fatigue (General disorders) | 16 (49) | 15 (29)
Anorexia (Gastrointestinal disorders) | 5 (10) | 4 (5)
Lymphocyte count decreased (Investigations) | 11 (49) | 13 (41)
Injection site reaction (Skin and subcutaneous tissue disorders) | 17 (114) | 3 (7)
Alanine aminotransaminase increased (Investigations) | 7 (15) | 9 (18)
Aspartate aminotransaminase increased (Investigations) | 9 (25) | 9 (19)
Alkaline phosphatase increased (Investigations) | 8 (14) | 4 (8)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4)
Blood bilirubin increased (Investigations) | 1 (2) | 4 (8)
CPK increased (Investigations) | 1 (1) | 0 (0)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (5) | 2 (6)
Cardiac disorders - Other, specify (tachycardia) (Cardiac disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 2 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 5 (7) | 8 (11)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (10) | 5 (7)
Creatinine increased (Investigations) | 3 (8) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 10 (23) | 9 (27)
Dizziness (Nervous system disorders) | 4 (16) | 2 (2)
Dry mouth (Gastrointestinal disorders) | 2 (3) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 (21) | 4 (5)
Edema face (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Edema limbs (Blood and lymphatic system disorders) | 10 (13) | 2 (2)
Gait disturbance (Musculoskeletal and connective tissue disorders) | 1 (3) | 0 (0)
Eyelid function disorder (Eye disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 5 (5) | 6 (13)
Flu-like syndrome (General disorders) | 3 (3) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 12 (45) | 13 (38)
Alopecia (Skin and subcutaneous tissue disorders) | 15 (18) | 13 (13)
Dyspepsia (Gastrointestinal disorders) | 1 (5) | 3 (3)
Hemoglobinuria (Renal and urinary disorders) | 2 (2) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (stomatitis) (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 1 (1) | 1 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0) — extravasation lt. forearm extravasation - infusion site lt. arm skin - annular quarter sized raised, red, uncomfortable at previous Denver insertion site
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 3 (4) | 3 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 3 (9) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (7) | 2 (4)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — muscle spasm, back, lt. foot/toe, jaw
Nail infection (Infections and infestations) | 1 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 10 (16) | 7 (21)
Neutrophil count decreased (Investigations) | 10 (39) | 6 (9)
Pain (General disorders) | 6 (9) | 2 (5)
Pruritis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (4)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 1 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (2) | 2 (2)
Allergic reaction (Immune system disorders) | 3 (4) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 14 (56) | 10 (43)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (6) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (6) | 1 (1)
Blood and lymphatic system disorders - Other, specify (hemoglobin, decreased) (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 2 (2)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 2 (5) | 1 (1)
Cholesterol high (Investigations) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 (9) | 4 (5)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 3 (9)
Platelet count decreased (Investigations) | 4 (7) | 2 (2)
Pericardial effusion (Cardiac disorders) | 4 (5) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 4 (6) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 4 (6)
Proteinuria (Renal and urinary disorders) | 5 (8) | 4 (4)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 6 (9) | 5 (12)
Sinus tachycardia (Cardiac disorders) | 2 (3) | 2 (4)
Dysgeusia (Gastrointestinal disorders) | 8 (9) | 4 (6)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Tremor (Nervous system disorders) | 2 (2) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperuricemia (Metabolism and nutrition disorders) | 3 (3) | 1 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (12) | 4 (7)
Watering eyes (Eye disorders) | 12 (15) | 9 (10)
Weight loss (Investigations) | 1 (2) | 1 (1)
Cardiac troponin I increased (Cardiac disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (8) | 1 (1)
Facial nerve disorder (Nervous system disorders) | 1 (1) | 1 (1)
Eye disorders - Other, specify (eye disorder: twitch; eye tearing) (Eye disorders) | 2 (2) | 0 (0)
General disorders and administration site conditions - Other, specify (General disorders) | 4 (5) | 0 (0) — body aches; decrease in taste; drowsiness; loss of taste; stomatitis
Mucositis oral (Gastrointestinal disorders) | 6 (7) | 4 (6)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (15) | 3 (9)
Hypoalbuminemia (Metabolism and nutrition disorders) | 14 (48) | 10 (32)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Infusion site extravasation (General disorders) | 1 (1) | 0 (0)
Investigations - Other, specify (elevated LDH) (Investigations) | 1 (7) | 0 (0)
Metabolism and nutrition disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (5) | 0 (0) — albumin decreased; BUN, decreased; bilirubin increased
CD4 lymphocytes decreased (Investigations) | 1 (1) | 1 (4)
Paronychia (Infections and infestations) | 1 (2) | 1 (1)
Surgical and medical procedures - Other, specify (surgical procedure, internal fixation) (Surgical and medical procedures) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 3 (4)
White blood cell decreased (Investigations) | 10 (59) | 11 (23)
Infections and infestations - Other, specify (left middle finger; port infection) (Infections and infestations) | 2 (2) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 3 (4) | 3 (3)
Nail loss (Skin and subcutaneous tissue disorders) | 6 (6) | 5 (5)
Nail ridging (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Nervous system disorders - Other, specify-neuropathy; neuropathy: toes; Rt finger tip numbness) (Nervous system disorders) | 5 (5) | 0 (0)
Non-cardiac chest pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
Palmer-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Paresthesia (Nervous system disorders) | 4 (5) | 5 (5)
Peripheral sensory neuropathy (Nervous system disorders) | 7 (14) | 6 (7)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (8) | 3 (4)
Sinusitis (Infections and infestations) | 1 (1) | 2 (2)
Skin induration (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Tooth infection (Infections and infestations) | 1 (1) | 0 (0)
Vascular disorders - Other, specify (Rt side eye; subconj. hem) (Vascular disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2)
Blood and lymphatic system disorders - Other, specify (anemia; hemoglobin decreased)) (Blood and lymphatic system disorders) | 0 (0) | 3 (5)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Eye disorders - Other, specify (eye tearing; eye tearing, watery eyes; eye redness)) (Eye disorders) | 0 (0) | 3 (3)
Fibrinogen decreased (Investigations) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (3)
General disorders and administration site conditions - Other, specify (General disorders) | 0 (0) | 3 (3) — stomatitis the patient had a cold
Hot flashes (Vascular disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 3 (6)
Infections and infestations - Other, specify (upper respiratiry infection) (Infections and infestations) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 2 (2)
Investigations - Other, specify (Investigations) | 0 (0) | 3 (6) — neutrophil count decreased; white blood cells decreased; BUN decreased 7mg/dL; bicarbonate, serum low; creatine kinase increased 22 mg/dl; lymphocyte count decreased
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 0 (0) | 3 (13) — albumin decreased; creatinine kinase decreased; creatinine decreased; creatine decreased; hemoglobin decreased; iron decreased; potassium decreased; sodium decreased; sodium increased; total protein, low
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Oral pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Reproductive system and breast disorders - Other, specify (dyspareunia) (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (rhinorrhea) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (8) — big toes and thumbs; general itching; peeling hands; rash (interior ankles); redden area at base of neck
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (4)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Weight gain (Investigations) | 0 (0) | 1 (2)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) — muscle spasm; musculoskeletal and connective tissue disorder - other, specify: toe cramp; myalgia/arthralgia (knee pain)
Palpitations (Cardiac disorders) | 2 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
The goal of this study was to get preliminary evidence of improved progression free survival with the combination compared with docetaxel alone and obtain data on which to plan a larger more definitive study in a more uniform patient population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No